CLINICAL TRIAL: NCT00555191
Title: Fructose Malabsorption in Northern Norway. Fructose Malabsorption and Irritable Bowel Syndrome.
Brief Title: Fructose Malabsorption in Northern Norway
Acronym: FINN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Nordlandssykehuset HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-136/2006(REK); 2006/136(REK-N) (Registry Identifier: Regional ethic comittee, REK-Nord); 15567/NSD (Other: Norsk samfinnsvitenskapelig datatjeneste); Ref 1204 Biobankregisteret (Registry Identifier: Biobankregisteret)
Record Dates: First submitted 2007-11-06; First posted 2007-11-08 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Irritable Bowel Syndrome; Fructose Malabsorption
Keywords: fructose; Irritable bowel syndrome; malabsorption; Glut5 transporter gene
MeSH Terms: conditions — Irritable Bowel Syndrome; Fructose Intolerance; Malabsorption Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): PATIENTS IN THIS ARM IS INSTRUCTED IN FRUCTOSE REDUCED DIET FOR A PERIOD OF 3 MONTHS
  Interventions: Behavioral: diet restriction
- 2 (No Intervention): these patients use their usual diet

INTERVENTIONS:
Behavioral: diet restriction — each meal should contain less than 2 gm fructose
  Arms: 1

SUMMARY:
Different published studies has shown a possible co-variation between leakage of fructose to the great bowel and exacerbation of irritable bowel syndrome (IBS) symptoms.

The aim of the FINN trial is to study the role of fructose malabsorption in patients with IBS in order to evaluate different diagnostic criteria for fructose malabsorption and at the same time study the effect of diet treatment in this cohort of patients and estimate the prevalence of fructose malabsorption.

ELIGIBILITY:
Inclusion Criteria:

* IBS patients satisfying ROME 2 diagnostic criteria

Exclusion Criteria:

* Seriously ill
* Organic abdominal disease
* Other functional bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2007-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
VAS score og specific abdominal complaints.SGA score of relief related to abdominal complaints. | 12 weeks

SECONDARY OUTCOMES:
Estimate sensitivity,specificity,negative and positive predictive value using 50 gm fructose in breath test.Validate questionary for intolerance.Validate VAS in judging changes in abdominal complaint.Examine polymorphism i Glut5 transporter gene. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jon Florholmen, MD PhD, Principal Investigator — University Hospital of North Norway, Department of Gastroenterology
Locations (1):
- Hospital of Rana Medical Dep. Helgelandsykehuset HF, Mo i Rana, Nordland, Norway

IPD SHARING:
Plan to Share IPD: Yes
Data already published in two articles published in Scandinavian Journal of Gastroenterology 2013 48: 936-943 DOI: 10.2109/00365521.2013.812139 andWorld Journal of Gastroenterology 2015 May 14;21(18) 5445-5754 DOI: 10.3748/ wjg.v21.i18.5677

REFERENCES:
- [Derived] Berg LK, Fagerli E, Myhre AO, Florholmen J, Goll R. Self-reported dietary fructose intolerance in irritable bowel syndrome: Proposed diagnostic criteria. World J Gastroenterol. 2015 May 14;21(18):5677-84. doi: 10.3748/wjg.v21.i18.5677. PMID 25987795